CLINICAL TRIAL: NCT02059941
Title: Managing Severe Traumatic Brain Injury (TBI) Without Intracranial Pressure Monitoring (ICP)- Guidelines Development and Testing
Brief Title: Managing Severe Traumatic Brain Injury (TBI) Without Intracranial Pressure Monitoring (ICP) Monitoring Guidelines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Randall M. Chesnut, Professor, Neurological Surgery, University of Washington
Other Study IDs: 44679
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Brain Injury
Keywords: Severe traumatic brain injury, ICP, Latin America, outcomes
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Management of intracranial hypertension (ICH) in patients with severe traumatic brain injury (sTBI) is crucial to their survival and optimal recovery. The evidence-based Guidelines for the Management of Severe Traumatic Brain Injury, 3rd Edition recommends use of intracranial pressure (ICP) monitors to assess ICH and guide intervention. Unfortunately, only a small percentage of the world has the resources and capability to routinely monitor ICP.

The objective of this proposal is to create and test guidelines for the treatment of severe TBI in the absence of ICP monitoring.

DETAILED DESCRIPTION:
Management of intracranial hypertension (ICH) in patients with severe traumatic brain injury (TBI) is crucial to their survival and optimal recovery. The evidence-based Guidelines for the Management of Severe Traumatic Brain Injury, 3rd Edition recommends use of intracranial pressure (ICP) monitors to assess ICH and know when and how to intervene. Unfortunately in most areas of the world there is no access to ICP monitor technology. This means that most people with severe TBI are treated without use of ICP monitoring. There are no Guidelines and no literature on how to treat severe TBI without use of ICP monitors.

The objective of this project is to create guidelines for the treatment of severe TBI in the absence of ICP monitoring and test them. We propose to derive these guidelines by working with a team of clinicians that practice in austere environments in low-to-middle income countries (LMICs) and routinely make decisions based either on a treatment protocol, their clinical experience, or both. We will use a new, systematic and innovative technology and process to accomplish consensus for the guidelines among the clinicians. We will implement the Consensus-Based Guidelines (CBG) in resource-poor centers, some of which have prior exposure to less well developed ad hoc protocols for treatment of TBI, and others that do not have prior exposure. We will test the influence of the CBG on outcomes of severe TBI in a before/after design in these two sets of centers. In the first two years, patients will be treated according to the ad hoc protocol or according to individual clinician best judgment. Then the Guidelines will be developed, all sites will be trained in their use, and they will be used to guide treatment in all sites for the next 2 years. .We will evaluate the effect of using an ad hoc protocol by comparing outcomes between the two sets of centers before the Guidelines are developed. In each set of centers we will evaluate the effect of using the consensus-based guideline protocol compared to either no protocol or the ad hoc protocol by comparing the outcomes in the first and second periods. Finally, we will evaluate how much more the consensus-based protocol effects outcome than the ad hoc protocol by comparing the difference from the first to the second period between the two sets of sites

In accomplishing the study objectives, we will create and test a guideline for the treatment of severe TBI that could be used globally to improve outcomes for these patients. We will validate in LMICs a new, systematic and innovative technology and process to accomplish consensus that was derived in an HIC. Finally, we will train personnel in centers new to research in how to conduct high-quality scientific studies, and will extend the training for the personnel with whom we have been working, solidifying previous capacity-building efforts, and initiating new efforts.

ELIGIBILITY:
Inclusion Criteria:

* Non-penetrating TBI
* Post-resuscitation Glasgow Coma Scale score (GCS) ≤ 8, and GCS Motor score ≤ 5, or Deterioration to those values within 48 hours of injury
* Age 13 years or older
* Consent to participate signed by Legally Authorized Representative (LAR)

Exclusion Criteria:

* GCS of 3 with bilateral fixed and dilated pupils and/or decision to not actively treat prior to enrolment into study
* Prisoner
* No consent
* Non-survivable injury
* Other (e.g., Pre-injury life expectancy under 1 year)
* Pre-existing neurological disability that would not allow follow-up

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study, there will be about 780 study subjects from 14 sites in Latin America. Subjects will be about 390 from clinical sites previously exposed to protocols for management of TBI, and about 390 from sites without prior exposure to protocols. Half of the study subjects (about 390 total) will be treated in accordance with a consensus-based protocol. Subjects will consist of patients with TBIs sufficiently severe to fulfill the inclusion criteria. To qualify, patients must be 13 or older and have a non-penetrating traumatic brain injury. The major criterion is severe TBI to be treated without the use of intracranial pressure monitoring
Sampling Method: Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2012-09-30 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The Galveston Orientation and Amnesia Test (GOAT | up to six months
  brief questionnaire that assesses orientation to time, place and person as well as post traumatic and retrograde amnesia. For this study, only the mental status portions of the measure will be used.
Color Trails Test | up to six months
  used to examine sustained and divided attention as well as mental flexibility. This is a two-part paper-pencil test measuring visual tracking. Part 1 requires the subject to connect 25 circles numbered 1 through 25, in sequence, distributed over a white sheet of paper, as quickly as possible. Part 2 is more complex and requires the person to connect the 25 numbered circles but alternating between pink and yellow colors. The scores obtained are the number of seconds required to complete each part of the test.
Spanish verbal learning test | up to six months
  consists of 16 words that the subject needs to learn over 5 trials with recall after each presentation. The score consists of the sum of correct recall over 5 trials. Delayed recall trial obtained 30 minutes later
Symbol Search subtest of the Wechsler Adult Intelligence | up to six months
  a measure of information processing speed. On this task the subject is presented with a pair of target symbols and must scan a search group of symbols to determine if there is a match.
The Glasgow Outcome Scale - Extended (GOSE) | up to six months
  score is obtained by a structured interview format that identifies specific criteria for assigning an outcome category. Outcome categories range from 1 (Dead) to 8 (Upper good recovery).
Functional Status Examination (FSE) | up to six months
  Outcome is examined in personal care, ambulation, mobility, major activities (i.e. work, school), home management, leisure and recreation, social integration, cognitive/behavioral competency and standard of living. These areas are evaluated using the concept of dependency to operationally define outcome at four levels. The first level signifies no change, the second level signifies difficulty in performing the activity although the person is still independent, the third level signifies dependence on others some of the time, and the fourth level signifies nonperformance or inability to perform the activity or total dependence on others.
Satisfaction with Life Scale (SWL) | up to six months
  a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time.
The Euroqol | up to six months
  is a standardized instrument to measure health outcome on 5 dimensions; Mobility, Self-Care, Usual Activities, Pain and Depression/Anxiety. It typically takes only a few minutes to complete.
Structured interview | up to six months
  is a questionnaire that obtains pre-injury demographic information (e.g., age, gender, nationality, race, ethnicity, education, medical history etc.) and pre- and post-injury information on marital status, employment history, living situation, and drug and alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Randall M Chesnut, MD, Principal Investigator — University of Washington
Locations (13):
- Bolivia (4):
  - Hospital Viedma, Cochabamba
  - Hospital Japones, Santa Cruz de la Sierra
  - Hospital San Juan de Dios, Santa Cruz de la Sierra
  - Hospital San Juan de Dios, Tarija
- Colombia (4):
  - Fundacion Clinica Campbell, Barranquilla
  - Clinica Universitaria Rafael Uribe, Cali
  - Hospital Erasmo Meoz #1, Cúcuta
  - Hospital Erasmo Meoz #2, Cúcuta
- Ecuador (2):
  - Hospital Jose Carrasco Arteaga, Cuenca
  - Hospital Espejo, Quito
- Venezuela (3):
  - Hospital Luis Razetti, Barcelona
  - Hospital Luis Razetti, Barinas
  - Hospital Dr. Patrocinio Penuela Ruiz, Cristobal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alali AS, Temkin N, Barber J, Pridgeon J, Chaddock K, Dikmen S, Hendrickson P, Videtta W, Lujan S, Petroni G, Guadagnoli N, Urbina Z, Chesnut RM. A clinical decision rule to predict intracranial hypertension in severe traumatic brain injury. J Neurosurg. 2018 Sep 28;131(2):612-619. doi: 10.3171/2018.4.JNS173166. Print 2019 Aug 1. PMID 30265194